CLINICAL TRIAL: NCT05057806
Title: Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors, Ketones, and Cardiovascular Benefit Research Plan
Brief Title: SGLT2 Inhibitors, Ketones, and Cardiovascular Benefit Research Plan
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Max and Minnie Tomerlin Voelcker Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC20210528H; 2021176 (Other Grant/Funding Number: Doris Duke Charitable Foundation)
Record Dates: First submitted 2021-09-15; First posted 2021-09-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Type2 Diabetes; Heart Failure With Preserved Ejection Fraction
Keywords: Ketones; Cardiovascular benefit
MeSH Terms: conditions — Ketosis | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: A randomized (2:1) placebo controlled double blind study
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin Group (Experimental): Subjects will be randomized 2:1 to receive empagliflozin, 25mg/day for 3 months
  Interventions: Drug: Empagliflozin 25 MG
- Placebo group (Placebo Comparator): Subjects will be randomized to receive the empagliflozin placebo for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Empagliflozin 25MG will be administered orally once per day for 3 months
  Other Names: Jardiance
  Arms: Empagliflozin Group
Drug: Placebo — The placebo will be administered orally once per day for 3 months
  Other Names: Placebo for Empagliflozin
  Arms: Placebo group

SUMMARY:
The study team will examine the effects of SGLT2i (and SGLT2i-induced increases in plasma ketone concentrations) on skeletal muscle and cardiac ketone uptake, skeletal muscle bioenergetics, cardiopulmonary exercise capacity, and patient-reported functional outcomes.

DETAILED DESCRIPTION:
The study team will examine effects of elevated plasma ketones caused by 12-week treatment with an SGLT2i (empagliflozin) treatment in participants with T2DM and HF. The study team will focus on three possible mechanisms of action for these effects and test the following:

(i) Skeletal muscle bioenergetics. Using 31P-MRS, the team will quantitate phosphocreatine [PCr], ATP, inorganic phosphate, phosphodiester, and intracellular pH. With 1H-MRS, and will measure intramyocellular lipid content at rest and ATPmax production after exercise. The team will examine the relationships between phosphorous metabolite concentrations, intramyocellular lipid content, and ATP generation before and after 12 weeks of SGLT2 inhibition.

(ii) Cardiopulmonary functional capacity.

(iii) Improvements in Patient-Reported Outcomes (PRO). The Patient-Reported Outcomes Measure Information System (PROMIS) Item Bank v2.0 - Physical Function - Short Form 20a will be used to evaluate self-reported physical function and well-being. This tool is a well-developed and validated method to obtain patient self-reported parameters of health in adults.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Class II-III New York Heart Association (NYHA) heart failure and reduced ejection fraction (EF) <50%
* Age 18-80 years
* BMI 23-38 kg/m2
* Glycated hemoglobin (HbA1c) 5.5-10%
* Blood Pressure (BP) ≤ 145/85 mmHg
* Estimated glomerular filtration rate (eGFR) ≥30 ml/min•1.73 m2
* Stable dose of guideline-directed medications for heart failure and Diabetes
* Stable body weight (±4 pounds) over the last 3 months
* Does not suffer from severe claustrophobia
* No contraindication for MRI (metal plates, screws, shrapnel, pins, or cardiac pacemaker)

Exclusion Criteria:

* Subjects treated with an SGLT2 inhibitor, a glucagon-like peptide-1 receptor agonist (GLP-1 RA) or pioglitazone
* Pregnancy, lactation or plans to become pregnant
* Allergy/sensitivity to study drugs or their ingredients
* Cancer
* Current drug or alcohol use or dependence
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Phosphocreatine | Baseline to 3 months
  A measure of phosphocreatine change from baseline to study end
Change in Adenosine Triphosphate (ATP) | Baseline to 3 months
  A measure of ATP change from baseline to study end
Change in Inorganic Phosphate | Baseline to 3 months
  A measure of inorganic phosphate change from baseline to study end
Change in Phosphodiester | Baseline to 3 months
  A measure of phosphodiester change from baseline to study end
ATPmax production | Baseline to 3 months
  Exercise induced ATPmax production change

SECONDARY OUTCOMES:
Plasma Beta-hydroxybutyrate (β-OH-B) | Baseline to 3 months
  Change in β-OH-B
Acetoacetate concentrations | Baseline to 3 months
  Change in acetoacetate concentrations
Cardiopulmonary Function | Baseline to 3 months
  Change in cardiopulmonary functional capacity using oxygen uptake (VO2)
6 minute walk test | Baseline to 3 months
  Change in the distance that can be covered in a 6 minute walk test
Patient-Reported Outcomes Measure Information System (PROMIS) | Baseline to 3 months
  Change in Physical function will be assessed by the PROMIS Item band v2.0 -Physical Function -Short Form 20a to evaluate patient-reported outcomes of physical function and well being.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Solis-Herrera, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (2):
- United States (2):
  - Texas Diabetes Institute - University Health System, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
The PI will actively participate in journal clubs and symposia and present abstracts at national meetings, as well as submitting manuscripts to top peer-reviewed journals.
Supporting Information: Study Protocol, SAP